CLINICAL TRIAL: NCT05220579
Title: A Randomized Blind Placebo-controlled 3rd Phase Study of the Safety and Efficacy of the Device "Device for Non-invasive Electromagnetic Therapy "TOR" in 236 Patients Diagnosed With Moderate Coronavirus Infection
Brief Title: Clinical Trial of a Medical Device "Device for Non-invasive Electromagnetic Therapy "TOR" in the Treatment of COVID-19"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concern GRANIT (Industry)
Collaborators: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SamaraTOR1
Record Dates: First submitted 2022-01-19; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infection COVID-19
Keywords: Coronavirus Infection; COVID-19; electromagnetic therapy; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled double-blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The "TOR" device was provided by the sponsor to the investigators with screened indicators on the front panel. The device was switched on / off by a medical monitor without the participation of medical personnel and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure to "TOR" device (Experimental): Patients undergo standard therapy + exposure to the "TOR" device
  Modes of patients' treatment with the "TOR" device:
  The exposure is carried out for at least 5 (five) days in a row for at least 4 hours daily in the 15 + 15 mode (15 minutes exposure + 15 minutes break).
  Standard therapy was prescribed in accordance with the recommended treatment regimens presented in the guidelines of the the Ministry of Health of Russia "Prevention, diagnosis and treatment of coronavirus infection (COVID-19) No. 9 dated 26.10. 2020)".
  Interventions: Device: Exposure to "TOR" device
- Control (No Intervention): Patients received standard therapy
  Standard therapy was prescribed in accordance with the recommended treatment regimens presented in the guidelines of the the Ministry of Health of Russia "Prevention, diagnosis and treatment of coronavirus infection (COVID-19) No. 9 dated 26.10. 2020)".
- Placebo (exposure to switched off "TOR" device) (Placebo Comparator): Patients undergo standard therapy + a switched off "TOR" device was installed in the wards
  Standard therapy was prescribed in accordance with the recommended treatment regimens presented in the guidelines of the the Ministry of Health of Russia "Prevention, diagnosis and treatment of coronavirus infection (COVID-19) No. 9 dated 26.10. 2020)".
  Interventions: Device: Exposure to switched off "TOR" device

INTERVENTIONS:
Device: Exposure to "TOR" device — Specific wave spectrum is directed by the "TOR" device to human tissues affected by the SARS-CoV-2 virus in order to disrupt its activity.
  Arms: Exposure to "TOR" device
Device: Exposure to switched off "TOR" device — The "TOR" device has screened indicators on the front panel. The device was switched on / off by a medical monitor without the participation of medical personnel and investigators.
  Arms: Placebo (exposure to switched off "TOR" device)

SUMMARY:
A clinical trial was conducted with human participation in order to assess the safety and efficacy of the medical device "TOR device for non-invasive electromagnetic therapy" when used as an adjunct in combination with standard COVID-19 treatment methods to accelerate the elimination (elimination) of the SARS-COV-2 virus from the nasopharynx in patients diagnosed with COVID-19.

Device principle of operation is based on the use of weak electromagnetic radiation, continuously induced by high-voltage pulses on the launcher of a pulsed electromagnetic field electrodes and causing noise in the SARS-CoV-2 virus.

The study included 236 patients who met all of the specified criteria: male and female patients aged ≥ 18 years with a coronavirus infection COVID-19 established diagnosis after specific testing, with a course of moderate disease, who do not require mechanical ventilation at the time of enrollment in the study. Infection with the SARS-CoV-2 virus had to be confirmed by PCR (nasopharyngeal and oropharyngeal swab). Informed consent was obtained from all patients. Results were statistically evaluated for 222 patients due to death and exclusion from the clinical study of 14 patients.

Patients of the test group were exposed to the "TOR" device for at least 5 (five) consecutive days for at least 4 hours daily in the 15 + 15 mode (15 minutes exposure + 15 minutes break) in combination with standard therapy. Patients in the placebo group were exposed to the switched off "TOR" device in combination with standard therapy. The control group received standard therapy. Standard therapy was prescribed in accordance with the recommended treatment regimens presented in the current version of the Temporary guidelines of the Ministry of Health of Russia "Prevention, diagnosis and treatment of coronavirus infection (COVID-19) No. 9 dated 26.10. 2020)". The study had the periods of screening (day 1, visit 0 - V0), treatment (days 2-6, visits 1-5 - V1-V5), discharge (day 7-14, visit 6 - V6), follow-up (day 26 -30, visit 7 - V7).

As a result of the clinical trial, it was established: "The device of non-invasive electromagnetic therapy "TOR" is safe when used as directed; effective as an adjuvant in combination with standard COVID-19 treatments to accelerate the elimination of the SARS-COV-2 virus from the nasopharynx.

DETAILED DESCRIPTION:
This is a research work with the participation of patients to study the effect of low-power electromagnetic radiation with a selected spectrum on infected cells and the SARS-CoV-2 virus itself.

In the course of work with wave emitters Research center of JSC "Concern GRANIT" conducted research in the field of the body's response to various wave frequencies and their combinations. In February 2020, the Concern's specialists, based on open information, created a computer model of the SARS-CoV-2 virus (COVID-19).

After creating the simulation, work was carried out to isolate the spectrum of the wave emanating from the COVID-19 virus colony and infected cells.

The resulting spectrum was modified for the purpose of noise pollution, and as a result the virus should lose activity and the standard line of behavior, which in turn should lead to a pause in its spread and enable the human immune system to cope with the infection on its own.

Based on these assumptions, the prepared wave spectrum was recorded into the "TOR" device emitter, acting with an electromagnetic field with an intensity not exceeding that of a household microwave oven.

The resulting spectrum is directed by the "TOR" device to human tissues affected by the SARS-CoV-2 virus in order to disrupt its activity.

Thus, investigators are talking about a method aimed to changing the SARS-CoV-2 virus behavior, both outside a healthy cell and inside an infected one.

The main task of this method is to bring low-power electromagnetic radiation with a selected spectrum as close as possible to infected cells and the virus itself.

The safety of the "TOR" device is confirmed by the Institute of the Federal State Budgetary Institution "ALL-RUSSIAN RESEARCH AND TESTING INSTITUTE OF MEDICAL TECHNOLOGY" of Roszdravnadzor (permission to conduct tests No. 876/2020 dated 10.12.2020 was issued by Roszdravnadzor).

The clinical study was carried out by the Federal State-Funded Educational Institution "Samara State Medical University" of the Ministry of Health of the Russian Federation.

Address: 443099 Samara region, Samara, st. Chapaevskaya, 89

The main objective of the study was: to assess the safety and efficacy of the medical device ""TOR" device for non-invasive electromagnetic therapy" when used as an adjunct in combination with standard COVID-19 treatment methods to accelerate the elimination (elimination) of the SARS-COV-2 virus from the nasopharynx in patients diagnosed with COVID-19.

Primary performance parameters were:

1. Dynamics of the SARS-CoV-2 virus replication activity (quantitative measurement of the genetic material of the virus (SARS-CoV-2 RNA) presence by PCR.
2. Dynamics of changes in the number of banded neutrophils.

Secondary performance parameters were:

1. Dynamics of saturation, respiratory rate.
2. The dynamics of changes in points on the WHO scale;
3. Dynamics of changes in points on the NEWS scale;

   Within the framework of the study, three cohorts were formed, in each patients were randomized into control group A, receiving only standard therapy, group B with the exposure to the "TOR" device plus standard therapy, and group C with simulated exposure to the "TOR" device (placebo) in combined with standard therapy. Patients were randomly assigned to groups by randomization at visit 1 (day 1) in a 1: 1 ratio. Group A consisted of 84 people (during the study, 73 patients remained due to the death of 11 patients), group B - 77 people (during the study, 75 patients remained due to the death of 2 patients), group C - 75 people (during the study 74 patients remained due to the death of 1 patient). Before the start of treatment, there were no statistically significant differences in the main clinical and functional parameters between patients of all groups, with the exception of anthropometric data, which was taken into account during the study.

   Cohort 1, exposure to the "TOR" device:

   • Patients undergo standard therapy + exposure to the "TOR" device

   Modes of patients' treatment with the "TOR" device:

   The exposure is carried out for at least 5 (five) days in a row for at least 4 hours daily in the 15 + 15 mode (15 minutes exposure + 15 minutes break).

   Longer exposure does not have a negative effect on the human body.

   Standard therapy was prescribed in accordance with the recommended treatment regimens presented in the guidelines of the the Ministry of Health of Russia "Prevention, diagnosis and treatment of coronavirus infection (COVID-19) No. 9 dated 26.10. 2020)".

   Cohort 2, placebo:

   • Patients undergo standard therapy + a switched off "TOR" device was installed in the wards

   Standard therapy was prescribed in accordance with the recommended treatment regimens presented in the guidelines of the the Ministry of Health of Russia "Prevention, diagnosis and treatment of coronavirus infection (COVID-19) No. 9 dated 26.10. 2020)".

   Cohort 3, control:

   • Patients received standard therapy

   Standard therapy was prescribed in accordance with the recommended treatment regimens presented in the guidelines of the the Ministry of Health of Russia "Prevention, diagnosis and treatment of coronavirus infection (COVID-19) No. 9 dated 26.10. 2020)".

   The study provides for the following periods:
   * Screening period / enrollment and initiation of symptomatic therapy - day 1, V0;
   * Treatment period - 2-6 days, V1-V5;
   * Discharge period - 7-14 days, V6;
   * Follow-up period: 26-30th day, V7. Thus, the maximum duration of participation in the study for one patient was 30 days.

   Visit 0 (screening / enrollment / initiation of symptomatic treatment): Day 1

   During the visit, the following procedures were performed:
   * Signing an informed consent form for participation in the study;
   * Collection of demographic data (date of birth, gender, age);
   * Collecting anamnesis;
   * Documenting a positive result of a PCR swab from the nasopharynx and / or oropharynx for SARS-CoV-2 no more than 72 hours old on the day of screening;
   * Documenting the results of a previously performed CT scan of the lungs;
   * Registration of complaints;
   * Registration of concomitant therapy;
   * Assessment of basic vital signs (blood pressure, heart rate [HR], respiratory rate) daily during hospitalization;
   * Measurement of axillary body temperature once a day
   * Physical examination;
   * Clinical blood test (hemoglobin level, hematocrit, erythrocyte count, leukocyte count, leukocyte count, platelet count, ESR);
   * Biochemical blood test (total protein, albumin, glucose, creatinine, urea, ALT, AST, total bilirubin, direct bilirubin, alkaline phosphatase, potassium, sodium, chlorine, C-reactive protein);
   * Coagulogram (activated partial thromboplastin time [APTT], PT, fibrinogen);
   * General urine analysis (color, transparency, relative density, pH, glucose, protein, ketone bodies, urobilinogen);
   * Assessment of SpO2 daily during hospitalization;
   * Electrocardiogram (ECG): performed to assess the QT interval;
   * Assessment of the condition according to the WHO scale;
   * Assessment of the condition according to the NEWS scale;
   * Assessment of inclusion / non-inclusion criteria;
   * Enrollment in the research;
   * Exposure of the method according to the Protocol;
   * Assessment of AEs / SAEs related to research procedures;
   * Assessment of exclusion criteria.

   Visits 1-5 (treatment period): days 2-6

   During the visit, the following procedures were performed:
   * Exposure of the patient with the "TOR" device;
   * Assessment of basic vital signs (blood pressure, heart rate, respiratory rate) daily during the period of hospitalization;
   * Daily measurement of axillary body temperature during hospitalization;
   * Assessment of SpO2 daily during hospitalization;
   * Assessment of the condition according to the WHO scale;
   * Assessment of the condition according to the NEWS scale;
   * Assessment of AE / SAE;
   * Assessment of exclusion criteria.

   Visit 6 (end of treatment period, discharge): Day 7-14

   During the visit, the following procedures were performed:
   * Assessment of basic vital signs (blood pressure, heart rate, respiratory rate);
   * Measurement of axillary body temperature;
   * Clinical blood test (hemoglobin level, hematocrit, erythrocyte count, leukocyte count, leukocyte count, platelet count, ESR);
   * Biochemical blood test (total protein, albumin, glucose, creatinine, urea, ALT, AST, total bilirubin, direct bilirubin, alkaline phosphatase, potassium, sodium, chlorine, C-reactive protein);
   * SpO2 assessment;
   * Assessment of the condition according to the WHO scale;
   * Assessment of the condition according to the NEWS scale;
   * Assessment of AE / SAE;
   * Assessment of exclusion criteria.

   Visit 7 (Follow-up): Day 26-30

   During the visit, the following procedures were performed:
   * Assessment of basic vital signs (blood pressure, heart rate, respiratory rate);
   * Measurement of axillary body temperature;
   * Clinical blood test (hemoglobin level, hematocrit, erythrocyte count, leukocyte count, leukocyte count, platelet count, ESR);
   * Biochemical blood test (total protein, albumin, glucose, creatinine, urea, ALT, AST, total bilirubin, direct bilirubin, alkaline phosphatase, potassium, sodium, chlorine, C-reactive protein);
   * SpO2 assessment;
   * Assessment of the condition according to the WHO scale;
   * Assessment of the condition according to the NEWS scale;
   * Assessment of AE / SAE.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 and over, diagnosed with coronavirus infection COVID-19 after specific testing. When the course of the disease progressed to a severe degree, patients were excluded from the study;
2. Signed consent to participate in the trial;
3. Patients hospitalized with COVID-19 disease. Positive result of a PCR test (biomaterial - a swab from the nasopharynx and / or oropharynx) for infection with the SARS-CoV-2 virus within 72 hours on the day of screening.
4. Patients with characteristic computed tomographic signs of the "ground-glass opacity" (one or two-sided spread) in combination with local foci of consolidation or without them;
5. Oxygen therapy is not required, or oxygen therapy is required using a face mask or nasal cannulas;
6. The duration of the disease from the first symptoms to the day of screening is not more than 7 days;
7. The ability to understand the requirements for research participants, to give written consent to participate in the research (including the use and transfer of information about the health of patients, relevant to the research) and to follow the procedures specified in the research protocol.

Exclusion Criteria:

1. The patient's desire to discontinue participation in the study (withdrawal of informed consent).
2. The decision of the investigating physician that the patient should be excluded for the benefit of the patient him/herself;
3. The patient refuses to cooperate with the investigator or is not disciplined;
4. Death of the patient;
5. Progressing of the disease to a severe degree.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
PCR | Day 5
  Dynamics of the SARS-CoV-2 virus replication activity (quantitative measurement of the genetic material of the virus (SARS-CoV-2 RNA) presence by PCR.
PCR | Day 14
  Dynamics of changes in the number of banded neutrophils.Dynamics of the SARS-CoV-2 virus replication activity (quantitative measurement of the genetic material of the virus (SARS-CoV-2 RNA) presence by PCR.
Banded neutrophils | Day 7
  Dynamics of changes in the number of banded neutrophils.
Banded neutrophils | Day 14
  Dynamics of changes in the number of banded neutrophils.
Banded neutrophils | Day 28
  Dynamics of changes in the number of banded neutrophils.

SECONDARY OUTCOMES:
Blood oxygen saturation | Day 2
  Dynamics of saturation.
Blood oxygen saturation | Day 3
  Dynamics of saturation.
Blood oxygen saturation | Day 4
  Dynamics of saturation.
Blood oxygen saturation | Day 5
  Dynamics of saturation.
Respiratory rate | Day 2
  Dynamics of respiratory rate.
Respiratory rate | Day 3
  Dynamics of respiratory rate.
Respiratory rate | Day 4
  Dynamics of respiratory rate.
Respiratory rate | Day 5
  Dynamics of respiratory rate.
Ordinal Scale for Clinical Improvement | Day 2
  The dynamics of changes in points on the scale (score 0-7, 0 - best outcome, 7 - worst outcome).
Ordinal Scale for Clinical Improvement | Day 3
  The dynamics of changes in points on the scale (score 0-7, 0 - best outcome, 7 - worst outcome).
Ordinal Scale for Clinical Improvement | Day 4
  The dynamics of changes in points on the scale (score 0-7, 0 - best outcome, 7 - worst outcome).
Ordinal Scale for Clinical Improvement | Day 5
  The dynamics of changes in points on the scale (score 0-7, 0 - best outcome, 7 - worst outcome).
Ordinal Scale for Clinical Improvement | Day 7
  The dynamics of changes in points on the scale (score 0-7, 0 - best outcome, 7 - worst outcome).
Ordinal Scale for Clinical Improvement | Day 14
  The dynamics of changes in points on the scale (score 0-7, 0 - best outcome, 7 - worst outcome).
Ordinal Scale for Clinical Improvement | Day 28
  The dynamics of changes in points on the scale (score 0-7, 0 - best outcome, 7 - worst outcome).
NEWS-2 (National Early Warning Score) scale | Day 2
  Dynamics of changes in points on the NEWS-2 scale (score 0 - >/= 7, 0 - best outcome, >/= 7 - worst outcome).
NEWS-2 (National Early Warning Score) scale | Day 3
  Dynamics of changes in points on the NEWS-2 scale (score 0 - >/= 7, 0 - best outcome, >/= 7 - worst outcome).
NEWS-2 (National Early Warning Score) scale | Day 4
  Dynamics of changes in points on the NEWS-2 scale (score 0 - >/= 7, 0 - best outcome, >/= 7 - worst outcome).
NEWS-2 (National Early Warning Score) scale | Day 5
  Dynamics of changes in points on the NEWS-2 scale (score 0 - >/= 7, 0 - best outcome, >/= 7 - worst outcome).
NEWS-2 (National Early Warning Score) scale | Day 7
  Dynamics of changes in points on the NEWS-2 scale (score 0 - >/= 7, 0 - best outcome, >/= 7 - worst outcome).
NEWS-2 (National Early Warning Score) scale | Day 14
  Dynamics of changes in points on the NEWS-2 scale (score 0 - >/= 7, 0 - best outcome, >/= 7 - worst outcome).
NEWS-2 (National Early Warning Score) scale | Day 28
  Dynamics of changes in points on the NEWS-2 scale (score 0 - >/= 7, 0 - best outcome, >/= 7 - worst outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Oleg V Fatenkov, Ph.D, M.D., Principal Investigator — Samara State Medical University
Locations (1):
- Concern GRANIT, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
We provide the Clinical Study Protocol upon request to the administrator's email.
Supporting Information: Study Protocol
Time Frame: Until December 31, 2022
Access Criteria: Upon request to the administrator's email address gryaznov.v@granit-concern.ru